CLINICAL TRIAL: NCT05223699
Title: A Phase I/II, Dose-Escalation Study of MGTA-117 in Patients With Adult Acute Myeloid Leukemia (AML) and Myelodysplasia-Excess Blasts (MDS-EB)
Brief Title: Study of MGTA-117 in Patients With Adult Acute Myeloid Leukemia (AML) and Myelodysplasia-Excess Blasts (MDS-EB)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Magenta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 117-HEM-101
Record Dates: First submitted 2022-01-14; First posted 2022-02-04 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplasia
Keywords: Acute Myeloid Leukemia; Myelodysplasia-Excess Blasts; MGTA-117; Hematopoietic stem cell transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single dose MGTA-117 (Experimental): Dosing of MGTA-117 prepared and administered by IV infusion.
  Interventions: Biological: MGTA-117

INTERVENTIONS:
Biological: MGTA-117 — MGTA-117 will be administered as an IV infusion

SUMMARY:
This research study is designed to selectively deplete CD117-positive cells from participants with AML and MDS-EB.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and potential anti-leukemia activity and to establish the minimum safe and biologically-effective dose of a single dose of MGTA-117 in relapsed/refractory (R/R) CD117+ AML participants and participants with MDS-EB. The study consists of escalating single-dose cohorts using a standard 3+3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a World Health Organization (WHO)-defined diagnosis of R/R AML and meet one of the following criteria:

   - The participant has experienced primary AML induction failure or R/R AML

   OR

   - The participant has a WHO-defined diagnosis of MDS-EB and has failed/is refractory to HMA

   OR

   - Presence of MRD in morphologic CR
2. CD117+ based on IHC or flow cytometry
3. Participant must have an identified HSC donor (related donor or unrelated donor), haplo-identical transplant donor, or umbilical blood donor.
4. Participant's Eastern Cooperative Oncology Group (ECOG) performance status must be ≤2.
5. Participant must have adequate baseline hepatic function. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤2 x upper limit of normal (ULN), and serum bilirubin ≤1.5 x ULN.
6. Estimated creatinine clearance ≥60 mL/min
7. Adequate cardiac function as demonstrated by cardiac left ventricular ejection fraction ≥40% or perform New York Heart Association (NYHA) classification I and II

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL).
2. Known active central nervous system (CNS) leukemia or chloroma (granulocyte sarcoma).
3. Received HSCT within 6 months prior to dosing
4. Received chimeric antigen-receptor cell therapies within 6 months prior to dosing
5. Has active graft-versus-host disease (GVHD).
6. Active hepatitis B (Hep-B) or hepatitis C (Hep-C) infection or history of human immunodeficiency virus (HIV).
7. Participant with a QTc value >470 msec
8. Participant has received another investigational drug or device within 14 days or 5 half-lives of dosing, whichever is longer.
9. Participant has any clinically significant medical condition, which in the opinion of the Investigator may place the participant at an unacceptable risk.
10. Active uncontrolled systemic bacterial, fungal, or viral infection
11. Participant has a history of serious allergic reactions, which in the opinion of the Investigator may pose an increased risk of serious infusion reactions.
12. Participant has had any systemic antileukemia treatment within 14 days except hydroxyurea, which is permitted until 24 hours prior to MGTA-117 dosing.
13. Participant has received prior anti-CD117 antibody treatment.
14. Participant has received gemtuzumab ozogamicin (Mylotarg) within the last 3 months prior to dosing.
15. Participant has received recent monoclonal antibody as anti-leukemic therapy within the last 30 days or 5 half-lives, whichever is longer.
16. Participant has received recent vaccination within the last 14 days prior to dosing.
17. Participant has Grade 2 or higher electrolyte abnormality at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence rate of treatment emergent adverse events (TEAEs) leading to study drug discontinuation | 21 days
Incidence rate of treatment emergent >= Grade 3 clinical laboratory abnormalities as assessed by CTCAE v5.0 | 21 days
Assess the clinically significant changes from baseline in vital signs, ECGs and laboratory parameters | 21 days
Pharmacokinetics profile of MGTA-117 | 21 days
  Investigate area under the curve (AUC)
Pharmacokinetics profile of MGTA-117 | 21 days
  Investigate maximum plasma concentration (Cmax)
Pharmacokinetics profile of MGTA-117 | 21 days
  Investigate time of maximum concentration (Tmax)
Pharmacokinetics profile of MGTA-117 | 21 days
  Investigate the half-life (t1/2)
Pharmacokinetics profile of MGTA-117 | 21 days
  Investigate the plasma concentration
To establish a minimum safe and biologically effective dose | 7 days
  Assess the CD117 receptor occupancy in circulating leukemic blasts
To establish a minimum safe and biologically effective dose | 21 days
  The incidence of qualifying protocol-defined dose-limiting toxicities

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - MD Anderson Cancer Center, Houston, Texas